CLINICAL TRIAL: NCT05609591
Title: Three Dietary Regimens in Pre-colonoscopic Bowel Preparation in Children : A Randomized Clinical Trial
Brief Title: Three Dietary Regimens in Pre-colonoscopic Bowel Preparation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FNF20210820
Record Dates: First submitted 2022-10-24; First posted 2022-11-08 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Bowel Preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liquid diet group (Experimental): From 8:00 on the day before colonoscopy, oral fluids including juice, rice soup, filtered vegetable juice/broth, lotus root powder and milk and egg soup were taken to ensure energy intake and blood glucose stability. The fasting starts at 9:00 AM on the day of colonoscopy.
  Interventions: Dietary Supplement: Liquid diet group
- Enteral nutrition group (Experimental): Oral administration of 100% short peptide enteral nutrition preparation from 8:00 on the day before colonoscopy. The fasting starts at 9:00 AM on the day of colonoscopy.
  Interventions: Dietary Supplement: Enteral nutrition group
- Low residual diet group (Experimental): From 8:00 on the day before colonoscopy, the patients were given oral administration of less residue food included gruel with grain only, peeled carrot, white gourd, powdered skin, tofu, vegetable, mud and fruit. The fasting starts at 9:00 AM on the day of colonoscopy.
  Interventions: Dietary Supplement: Low residual diet group

INTERVENTIONS:
Dietary Supplement: Liquid diet group — Fluid diet including juice, rice soup, filtered vegetable juice/broth, lotus root powder and milk and egg soup were given to children for bowel preparation.
  Arms: Liquid diet group
Dietary Supplement: Enteral nutrition group — 100% short peptide enteral nutrition are given to children for bowel preparation
  Arms: Enteral nutrition group
Dietary Supplement: Low residual diet group — Low residua diet included gruel with grain only, peeled carrot, white gourd, powdered skin, tofu, vegetable, mud and fruit. were given to children for bowel preparation
  Arms: Low residual diet group

SUMMARY:
To describe the feasibility and effectiveness of three dietary regimens in precolonoscopy bowel preparation in children

DETAILED DESCRIPTION:
The accuracy of endoscopic diagnosis and treatment of safety depends largely on the intestinal cleaning quality. Qualified bowel preparation is a prerequisite for clear vision during colonoscopy. Presently, the common diet for children before colonoscopy in China is a liquid or low residual diet. The liquid and low residual diet often have poor taste and satiety, often resulting in poor compliance of children, especially young children, who are often unwilling to eat a liquid diet, resulting in insufficient caloric supply and unstable blood glucose during bowel preparation. Enteral formula as a kind of high-energy and low-fiber diet has been applied in clinical practice. Currently, there is no comparison between liquid diet, low-residue diet, and enteral formulas in children's bowel preparation in China. Dietary restriction is an indispensable part to ensure the success of the bowel preparation program. There is an urgent need to conduct research on the application of various dietary programs in children's bowel preparation before colonoscopy in China. In order to provide high-quality evidence for the bowel preparation diet program for children.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 years～18 years old
2. Children under anesthesia for elective colonoscopy with bowel preparation

Exclusion Criteria:

1. Children who are unable to perform bowel preparation with polyethylene glycol-4000
2. Children whose guardians refuse to participate in this study
3. Children who are unable to eat orally
4. Children with stomy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 900 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale score | After the children finish their bowel preparation, an average of 5 minutes
  The nurse will use the Boston Bowel Preparation Scale colonoscopic to evaluate the intestinal fecal trait under colonoscope and record in the case report form. The right side (cecum and ascending colon), transverse colon (hepatic flexion and splenic flexion) and left side (descending colon, sigmoid colon and rectum) were scored respectively. 0 score: a large amount of solid stool remains in the colon; 1 score: liquid and semi-solid feces exist in some intestinal segments; 2 points: a small amount of feces remains, but does not affect the colonoscopic field of view; 3 points: no solid liquid fecal residue in the colon.
  The total score of the scale is 9 points, 8-9 points is excellent; 6-7 points is good; 4-5 points is average; 0-3 points is Poor.

SECONDARY OUTCOMES:
Revised-Bristol Stool Form Scale score | After the children finish their bowel preparation, an average of 5 minutes.
  The fecal traits are recorded in the case report form by the nurse with a Revised-Bristol Stool Form Scale according to the stool characteristics of children. The score was 8 points in order: 8 points: clear water stool, no residue; 7 points: turbid water sample, with or without a small amount of fecal residue; 6 points: velvet, unclear edge, mushy stool; 5 points: soft mass, clear edge; 4 points: like sausage or snake, smooth and soft; 3 points: sausage-shaped, but with cracks on the surface; 2 points: sausage-shaped, but in chunks; 1 point: scattered hard pieces, like nuts. A score of 8 indicates that the naked eye assessment of bowel preparation is qualified, and colonoscopy can be performed directly. A score of 6-7 indicates that bowel preparation is not sufficient, and a colonoscopy should be performed at the selected day. ≤5 points is recommended to cancel the colonoscopy on the same day and extend the bowel preparation time.
The times of enema | After the children finish their enema, an average of 1 minute.
  Children with substandard bowel preparation before colonoscopy were going to undergo enemas to ensure the visual clarity of colonoscopy. The times of enema will be recorded by the nurse who perform the enema in the case report form.
Number of defecation during bowel preparation | After the children finish their bowel preparation, an average of 1 minute.
  The number of defecation during bowel preparation will be recorded in the case report form by the nurse.
Medication compliance | After the children finish their bowel preparation, an average of 3 minutes.
  Children who complete less than 30% polyethylene glycol 4000 (PEG-4000) are defined as having poor compliance, completing 30%~60% PEG-4000 is fair compliance, completing 60%~80% PEG-4000 is good compliance, and great than 80% PEG-4000 is excellent compliance. The nurse will evaluate children's compliance according to their completion of PEG-4000 and record it in the case report form.
Adverse reactions of bowel preparation | During children's bowel preparation, an average of 24 hours.
  Acceptable safety indicators: occasional and mild nausea, vomiting, abdominal pain, abdominal distension; a few sporadic rashes; perianal discomfort.
  Indicators need to be closely monitored: frequent and severe vomiting, abdominal pain, abdominal distension, blood in the stool; Widespread or diffuse rash.
  Unacceptable indicators: fecal incontinence, dehydration, and electrolyte disturbance; intestinal perforation; shock.
  All the adverse reactions will be observed and recorded in the case report form by the nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gu, 3, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children'S Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
we will not make individual participant data available to other reseasrchers

REFERENCES:
- [Result] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Result] Belsey J, Epstein O, Heresbach D. Systematic review: oral bowel preparation for colonoscopy. Aliment Pharmacol Ther. 2007 Feb 15;25(4):373-84. doi: 10.1111/j.1365-2036.2006.03212.x. PMID 17269992
- [Result] Barkun A, Chiba N, Enns R, Marcon M, Natsheh S, Pham C, Sadowski D, Vanner S. Commonly used preparations for colonoscopy: efficacy, tolerability, and safety--a Canadian Association of Gastroenterology position paper. Can J Gastroenterol. 2006 Nov;20(11):699-710. doi: 10.1155/2006/915368. PMID 17111052
- [Result] Mytyk A, Lazowska-Przeorek I, Karolewska-Bochenek K, Kakol D, Banasiuk M, Walkowiak J, Albrecht P, Banaszkiewicz A. Clear Liquid Versus Low-fibre Diet in Bowel Cleansing for Colonoscopy in Children: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2018 May;66(5):720-724. doi: 10.1097/MPG.0000000000001832. PMID 29112090
- [Result] Wu R, Ji WY, Yang C, Zhan Q. A Systematic Review and Meta-Analysis of Low-Residue Diet Versus Clear Liquid Diet: Which Is Better for Bowel Preparation Before Colonoscopy? Gastroenterol Nurs. 2021 Sep-Oct 01;44(5):341-352. doi: 10.1097/SGA.0000000000000554. PMID 34238885